CLINICAL TRIAL: NCT06173986
Title: A Phase I/II Multicenter Study Evaluating the Efficacy and Safety of Induction Immunochemotherapy Followed by Concurrent Immuno-Chemoradiotherapy in Unresectable Locally Advanced Esophageal Squamous Cell Cancer(SCR-ESCC-02)
Brief Title: Immunotherapy in Combination With Chemoradiotherapy in Unresectable Locally Advanced Esophageal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Wen Yu, Vice Director of Radiation Oncology Department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCR-ESCC-02
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Unresectable Locally Advanced Esophageal Cancer
Keywords: Immunotherapy; Induction immunochemotherapy; Concurrent Immuno-Chemoradiotherapy; Unresectable locally advanced esophageal cancer; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Immunotherapy; 130-nm albumin-bound paclitaxel; Cisplatin; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IC+ICRT group (Experimental): 2 cycles of PD-1 inhibitor + nab-paclitaxel + cisplatin followed by concurrent PD-1 inhibitor + radiotherapy (45-50Gy/25fx) + nab-paclitaxel + cisplatin
  Interventions: Drug: PD-1inhibitor; Drug: nab-paclitaxel + cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: PD-1inhibitor — PD-1 inhibitor, Q3W, until disease progression or unacceptable toxicity or treatment reaches 1 year
  Other Names: Immunotherapy
Drug: nab-paclitaxel + cisplatin — Induction phase: nab-paclitaxel + cisplatin, Q3W × 2 cycles; Concurrent ICRT phase: nab-paclitaxel + cisplatin, QW × 5 cycles
  Other Names: Chemotherapy
Radiation: Radiotherapy — Primary tumor and metastatic lymph nodes, DT:45-50Gy/25fx, starting within 4 weeks following the completion of the last induction immunochemotherapy cycle

SUMMARY:
SCR-ESCC-02 is a multicenter, phase I/II clinical study to investigate the safety and efficacy of induction immunochemotherapy followed by concurrent chemoradiotherapy with anti-PD-1 therapy in patients diagnosed with locally advanced, unresectable esophageal cancer.

DETAILED DESCRIPTION:
Immunotherapy has shown promising results in advanced esophageal cancer, but its optimal integration into the management of unresectable locally advanced disease remains uncertain. The significant tumor regression and reduced tumor residual achieved through immunochemotherapy offer an opportunity to enhance the effectiveness of subsequent radiotherapy. This phase I/II clinical study aims to investigate the efficacy and safety of induction immunochemotherapy followed by concurrent chemoradiotherapy with anti-PD-1 for patients with unresectable locally advanced esophageal cancer. The study's co-primary endpoints are progression-free survival (PFS) and treatment completion rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
3. Clinical stage meeting the criteria of T1N+M0 or T2-4aN0-3M0 based on the 8th UICC-TNM classification.
4. Ineligibility for surgical resections due to patients' unwillingness for surgery, technically unresectable disease, or being medically unfit for surgery.
5. No prior anti-tumor treatment, including surgery, radiotherapy, chemotherapy, immunotherapy, or targeted therapy.
6. Adequate hematological, pulmonary, cardiac, hepatic, renal, and thyroid function.
7. Willingness to use contraception with an adequate method throughout the study.
8. Documented informed consent.

Exclusion Criteria:

1. History of malignant disease within the 5 years preceding enrollment or presence of other malignant tumors or non-squamous cell carcinoma components.
2. High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation as determined by the investigators.
3. Weight loss exceeding 20% within the 90 days prior to the first day of drug administration.
4. Presence of long-standing unhealed wounds or fractures or undergoing major surgical resections within 60 days preceding the first day of drug administration.
5. Presence of any severe or uncontrolled coexisting diseases, including but not limited to:

   * Uncontrolled hypertension
   * History of interstitial lung disease or non-infectious pneumonia
   * Active hepatitis B or C, syphilis, or other active and uncontrolled infections
   * Cardiac insufficiency (NYHA≥2)
   * Renal dysfunction requiring dialysis
   * Active autoimmune disease
   * History of acquired or congenital immunodeficiency diseases
6. Occurrence of serious arterial/venous thrombotic events within 6 months prior to the first day of drug administration.
7. History of psychotropic substance abuse or inability to quit, or patients with psychotic disorders.
8. Allergy to study drugs.
9. Patients deemed unsuitable for participation due to severe comorbidities or other reasons determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Assessed up to 60 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
Treatment completion rate | 1 year
  The Treatment Completion Rate is defined as the percentage of patients who successfully completed concurrent immuno-chemoradiotherapy.

SECONDARY OUTCOMES:
Objective response rate | 1 year
  Objective response rate (ORR), defined as the proportion of patients with a complete response or partial response after Immuno-Chemoradiotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST)
Overall survival | Assessed up to 60 months
  From date of randomization until the date of death from any cause
Incidence of Adverse events (AE) or severe adverse events (SAE) | 1 year
  Adverse events (AE) or severe adverse events (SAE) occurring within 3 months post-radiotherapy, and the incidence of treatment discontinuation due to AE/SAE

CONTACTS AND LOCATIONS:
Overall Officials: Wen Yu, M.D, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hulshof MCCM, Geijsen ED, Rozema T, Oppedijk V, Buijsen J, Neelis KJ, Nuyttens JJME, van der Sangen MJC, Jeene PM, Reinders JG, van Berge Henegouwen MI, Thano A, van Hooft JE, van Laarhoven HWM, van der Gaast A. Randomized Study on Dose Escalation in Definitive Chemoradiation for Patients With Locally Advanced Esophageal Cancer (ARTDECO Study). J Clin Oncol. 2021 Sep 1;39(25):2816-2824. doi: 10.1200/JCO.20.03697. Epub 2021 Jun 8. PMID 34101496
- [Background] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Background] Li C, Zhao S, Zheng Y, Han Y, Chen X, Cheng Z, Wu Y, Feng X, Qi W, Chen K, Xiang J, Li J, Lerut T, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for oesophageal squamous cell carcinoma (PALACE-1). Eur J Cancer. 2021 Feb;144:232-241. doi: 10.1016/j.ejca.2020.11.039. Epub 2020 Dec 26. PMID 33373868
- [Background] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Background] Shah MA, Bennouna J, Doi T, Shen L, Kato K, Adenis A, Mamon HJ, Moehler M, Fu X, Cho BC, Bordia S, Bhagia P, Shih CS, Desai A, Enzinger P. KEYNOTE-975 study design: a Phase III study of definitive chemoradiotherapy plus pembrolizumab in patients with esophageal carcinoma. Future Oncol. 2021 Apr;17(10):1143-1153. doi: 10.2217/fon-2020-0969. Epub 2021 Feb 3. PMID 33533655
- [Background] Yu R, Wang W, Li T, Li J, Zhao K, Wang W, Liang L, Wu H, Ai T, Huang W, Li L, Yu W, Wei C, Wang Y, Shen W, Xiao Z. RATIONALE 311: tislelizumab plus concurrent chemoradiotherapy for localized esophageal squamous cell carcinoma. Future Oncol. 2021 Nov;17(31):4081-4089. doi: 10.2217/fon-2021-0632. Epub 2021 Jul 16. PMID 34269067
- [Background] Wang Z, Shao C, Wang Y, Duan H, Pan M, Zhao J, Wang J, Ma Z, Li X, Yan X. Efficacy and safety of neoadjuvant immunotherapy in surgically resectable esophageal cancer: A systematic review and meta-analysis. Int J Surg. 2022 Aug;104:106767. doi: 10.1016/j.ijsu.2022.106767. Epub 2022 Jul 14. PMID 35840049
- [Background] Spigel DR, Faivre-Finn C, Gray JE, Vicente D, Planchard D, Paz-Ares L, Vansteenkiste JF, Garassino MC, Hui R, Quantin X, Rimner A, Wu YL, Ozguroglu M, Lee KH, Kato T, de Wit M, Kurata T, Reck M, Cho BC, Senan S, Naidoo J, Mann H, Newton M, Thiyagarajah P, Antonia SJ. Five-Year Survival Outcomes From the PACIFIC Trial: Durvalumab After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Apr 20;40(12):1301-1311. doi: 10.1200/JCO.21.01308. Epub 2022 Feb 2. PMID 35108059
- [Background] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008